CLINICAL TRIAL: NCT02940782
Title: Assessment of Postoperative Pain After Using Reciroc Versus One Shape NiTi Systems in Patients With Symptomatic Irreversible Pulpitis (A Randomized Clinical Trial): Part Two
Brief Title: Comparison Between Reciproc and Oneshape Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Abdullah Ali Soliman, Masters Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: reciproc_oneshape
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reciproc single file system (Experimental): It is a reciprocating NiTi file used for instrumentation of root canals in endodontic treatment
  Interventions: Procedure: Reciproc single file system; Device: X-smart Plus, Dentsply Maillefer, Ballaigues, Switzerland
- One Shape single file system (Active Comparator): It is a rotary NiTi file used for instrumentation of root canals in endodontic treatment
  Interventions: Procedure: One Shape single file system; Device: X-smart Plus, Dentsply Maillefer, Ballaigues, Switzerland

INTERVENTIONS:
Procedure: Reciproc single file system — A reciprocating Nickel Titanium single file system used for instrumentation of root canals in endodontic treatment.
  Arms: Reciproc single file system
Procedure: One Shape single file system — A rotary Nickel Titanium single file system used for instrumentation of root canals in endodontic treatment.
  Arms: One Shape single file system
Device: X-smart Plus, Dentsply Maillefer, Ballaigues, Switzerland — It is a micro-motor designed for performing root canal treatments with the reciprocating, single file technique or traditional continuous rotation file system.

SUMMARY:
A randomized clinical trial to assess postoperative pain in patients with symptomatic irreversible pulpitis after using Reciproc versus One Shape rotary NiTi Systems.

DETAILED DESCRIPTION:
The study aims at comparing postoperative pain after using two single-file NiTi systems, Reciproc reciprocating system and One Shape rotary system, for root canal instrumentation in patients with symptomatic irreversible pulpitis.

After the patient is found eligible, he/she will be randomly assigned to either the control (One Shape) or experimental group (Reciproc) and will be treated in a single visit.

Sequence of Procedural Steps:

1. Assessment of preoperative pain by NRS before administration of anesthesia.
2. Administration of local anesthesia using 2% lidocaine (1:100,000 adrenaline).
3. An access cavity will be done using a round bur and Endo-Z bur.
4. Isolation of the affected tooth with rubber dam.
5. Determination of the working length using an electronic apex locator, and confirmed by a radiograph using K-file. Then, the working length will be established at 0.5 mm up to the radiographic apex.
6. Canals will be explored with hand K-file ISO sizes 10, 15, 20.
7. Mechanical preparation for both groups will be as follows:

   * Experimental group:

     * Canals will be instrumented using Reciproc reciprocating system set on an electric motor, with adjusted torque and speed according to the manufacturer's instructions.
     * There is no need for coronal preflaring with a Gates Glidden drill or an orifice opener since the design of the Reciproc instrument allows any obstructions in the coronal third to be removed, as claimed by the manufacturer.
     * Reciproc file selection: R40 (40/0.06)
   * Control group:

     * Coronal preflaring will be performed using Gates Glidden drill.
     * Canals will be instrumented using One Shape single-file (25/0.06) set on an electric motor with adjusted torque and speed according to the manufacturer's instructions.
     * For wide canals, One Shape Apical (30/0.06, 37/0.06) will be used.
8. The rotary files will be introduced inside the canal using EDTA gel.
9. Canals will be irrigated with 2.6% sodium hypochlorite solution between every subsequent instrument. It is prepared by adding 10 ml of sterile distilled water to 10 ml of 5.25% sodium hypochlorite solution using a 27 gauge needle fit to 5ml disposable plastic syringe placed in the canal space without binding.
10. Canals will be dried with sterile paper points and obturated using lateral condensation technique. A spreader will be used to allow space for auxiliary cones, with resin-based root canal sealer.
11. The tooth will be sealed by temporary restoration, and postoperative pain will be assessed immediately after the end of treatment.
12. The patient will be phone called for follow up after 6, 12, 24, 48 and 72 hours.
13. The patient will be instructed to return to complete the treatment procedures until placing a full-coverage restoration.
14. The patient will be instructed to take one tablet 600 mg Ibuprofen if he/she experiences severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular premolar teeth with:

  * Single canal
  * Preoperative sharp pain.
  * Vital response of pulp tissue.
  * Normal periapical radiographic appearance or slight widening in lamina dura.
* Final diagnosis for an eligible patient will take place by radiograph and pulp testing.

Exclusion Criteria:

* Patients who have already consumed preoperative medication, such as analgesic, non-steroidal or steroidal anti-inflammatory drugs, within 12 hours before treatment.
* Patients who have more than one tooth in the same quadrant and/or opposite quadrant that require an endodontic treatment.
* Pregnant females.
* Patients having significant systemic disorder.
* If antibiotics have been administrated during the past two weeks preoperatively.
* Patients having bruxism or clenching.
* Teeth that have:

  * Non-vital pulp tissues.
  * Association with swelling or fistulous tract.
  * A pocket depth greater than 5 mm.
  * Previous endodontic treatment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the change in postoperative pain measured by the Numerical Rating Scale (0-10) | Immediately after treatment, then 6 hours, 12 hours, 24 hours and 72 hours after treatment.
  Pain intensity after root canal treatment will be measured using Numerical Rating Scale (0-10)

SECONDARY OUTCOMES:
Number of analgesics taken by the patient | 72 hours from the end of the endodontic treatment
  It will be recorded by the patient with time intervals

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Soliman, B.D.S, Principal Investigator — Faculty of Oral and Dental Medicine, Cairo University; Angie G Ghoneim, Study Director — Faculty of Oral and Dental Medicine, Cairo University; Shaimaa I Gawdat, Study Chair — Faculty of Oral and Dental Medicine, Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neelakantan P, Sharma S. Pain after single-visit root canal treatment with two single-file systems based on different kinematics--a prospective randomized multicenter clinical study. Clin Oral Investig. 2015 Dec;19(9):2211-7. doi: 10.1007/s00784-015-1448-x. Epub 2015 Mar 15. PMID 25773449
- [Background] Kherlakian D, Cunha RS, Ehrhardt IC, Zuolo ML, Kishen A, da Silveira Bueno CE. Comparison of the Incidence of Postoperative Pain after Using 2 Reciprocating Systems and a Continuous Rotary System: A Prospective Randomized Clinical Trial. J Endod. 2016 Feb;42(2):171-6. doi: 10.1016/j.joen.2015.10.011. Epub 2015 Nov 29. PMID 26614017